CLINICAL TRIAL: NCT02243904
Title: Study for Promotion of Health in Recycling Lead
Acronym: SPHERL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Jan A. Staessen, Professor of Medicine, KU Leuven
Other Study IDs: SPHERL
Record Dates: First submitted 2014-09-10; First posted 2014-09-18 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Occupational Exposure
Keywords: Autonomic nervous function; Blood pressure; Cardiovascular regulation; Lead; Occupational exposure; Renal function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lead exposure

SUMMARY:
Study for Promotion of Health in Recycling Lead (SPHERL) is a prospective 2-year follow-up study of lead workers with exposure levels varying between and within individuals. SPHERL addresses to what extent between-subject differences or within-subject changes in lead exposure may have a measurable impact on blood pressure, the cardiovascular system, renal function, the autonomic nervous system, peripheral nervous conduction velocity, and neurocognitive function.

At the beginning of December 2015, 70 participants were included in the study.

DETAILED DESCRIPTION:
Background

* Whether low-level lead exposure impacts on blood pressure, regulation of the cardiovascular system, glomerular or tubular renal function, sympathetic nervous modulation, peripheral nervous conduction velocity, and neurocognitive function remains uncertain.

Study Population

* SPHERL will enroll 500 lead recycling workers with changing lead exposure, who will be examined at baseline (2014-2015) and followed up at annual intervals for 2 years (2016-2017).

Methods

* Volunteers eligible for the study are (i) new and existing hires without previous occupational lead exposure who will be performing tasks with or without occupational lead exposure and (ii) existing hires with occupational lead exposure who will be transitioning to job tasks without occupational lead exposure within the next 2 years.
* Blood lead concentration will be the main biomarker of exposure.
* The main outcome variables are (i) blood pressure measured conventionally and by ambulatory monitoring, and analyzed as continuous or categorical variable, both cross-sectionally and longitudinally; (ii) indexes of glomerular and tubular renal function, (iii) heart rate variability analyzed in the frequency domain as measure of autonomous sympathetic modulation, (iv) peripheral nerve conductivity, (v) neurocognitive performance, (vi) and quality of life [the EuroQOL five dimensions (EQ-5D) questionnaire].

Expected Outcomes

* Assuming a 4-fold or higher surge in the blood lead concentration, the study is powered to demonstrate over 2 years an acceleration in the age-related rise of systolic blood pressure by 1 to 4 mm Hg or an increase of the coefficient of multiple determination (R2) from 0.22 to 0.24 by adding the change in the blood lead concentration to models relating changes in blood pressure to three other covariables. The longitudinal design of our study complies with the temporality principle of the Bradford-Hill criteria for assessing possible causality between outcomes and exposure.

ELIGIBILITY:
Inclusion Criteria:

* Women and men are eligible.
* New hires without previous occupational lead exposure who will be performing tasks with lead exposure or current employees without previous occupational lead exposure moving to tasks with exposure.
* Informed written consent.

Exclusion Criteria:

* Pregnancy.
* Any serious health condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited among the work force employed at lead recycling plants in North America.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2015-08; Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Annual change in systolic blood pressure as measured by 24-h ambulatory monitoring | Baseline, 1 year and 2 years

SECONDARY OUTCOMES:
Annual change in central hemodynamics | Baseline, 1 year and 2 years
  Annual changes in the central hemodynamics, including aortic blood pressure, the central systolic augmentation index, and aortic pulse wave velocity
Annual change in heart function | Baseline, 1 year and 2 years
  Annual changes in ECG-derived indexes
Annual change in renal function | Baseline, 1 year and 2 years
  Annual changes in glomerular and tubular renal function measured on a continuous scale and the incidence of renal dysfunction
Annual change in autonomic nervous function | Baseline, 1 year and 2 years
  Annual changes in alterations in the autonomic nervous cardiovascular modulation, as assessed by heart rate variability
Annual change in peripheral nervous conduction velocity | Baseline, 1 year and 2 years
  Annual changes in nerve conduction velocity
Annual change in neurocognitive performance | Baseline, 1 year and 2 years
  Annual changes in neurocognitive testing
Annual change in quality of life | Baseline, 1 year and 2 years
  Annual changes in self-assessed quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Staessen, MD, PhD, Principal Investigator — University of Leuven
Locations (1):
- University of Leuven, Leuven, Belgium

REFERENCES:
- [Result] Hara A, Gu YM, Petit T, Liu YP, Jacobs L, Zhang ZY, Yang WY, Jin Y, Thijs L, Wei FF, Nawrot TS, Staessen JA. Study for Promotion of Health in Recycling Lead - Rationale and design. Blood Press. 2015 Jun;24(3):147-57. doi: 10.3109/08037051.2014.996409. Epub 2015 Jan 26. PMID 25620211
- [Derived] Yu YL, An DW, Yang WY, Verhamme P, Allegaert K, Nawrot TS, Staessen JA. Blood pressure and renal function responses in workers exposed to lead for up to six years. J Clin Hypertens (Greenwich). 2023 Dec;25(12):1086-1095. doi: 10.1111/jch.14748. Epub 2023 Nov 8. PMID 37938055
- [Derived] Yu YL, Thijs L, Saenen N, Melgarejo JD, Wei DM, Yang WY, Yu CG, Roels HA, Nawrot TS, Maestre GE, Staessen JA, Zhang ZY. Two-year neurocognitive responses to first occupational lead exposure. Scand J Work Environ Health. 2021 Apr 1;47(3):233-243. doi: 10.5271/sjweh.3940. Epub 2020 Dec 4. PMID 33274751
- [Derived] Yu YL, Yang WY, Thijs L, Melgarejo JD, Yu CG, Wei DM, Wei FF, Nawrot TS, Zhang ZY, Staessen JA. Two-Year Responses of Office and Ambulatory Blood Pressure to First Occupational Lead Exposure. Hypertension. 2020 Oct;76(4):1299-1307. doi: 10.1161/HYPERTENSIONAHA.120.15590. Epub 2020 Sep 9. PMID 32903104
- [Derived] Yu CG, Wei FF, Yang WY, Zhang ZY, Mujaj B, Thijs L, Feng YM, Staessen JA. Heart rate variability and peripheral nerve conduction velocity in relation to blood lead in newly hired lead workers. Occup Environ Med. 2019 Jun;76(6):382-388. doi: 10.1136/oemed-2018-105379. Epub 2019 Mar 30. PMID 30928907